CLINICAL TRIAL: NCT05761106
Title: Effect of Exercises on Convergence Insufficiency in Individuals With Temporomandibular Disorders: Clinical, Randomized, Blinded Trial
Brief Title: Effect of Exercises on Convergence Insufficiency in Individuals With Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Convergence Insufficiency
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Convergence Insufficiency
Keywords: Convergence Insufficiency; Temporomandibular Disorder; Clinical trials; oculomotor therapy; Physiotherapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Ocular Motility Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two researchers will be part of the protocol.One will be responsible for pre and post intervention assessments and will be blind to the type of interventionThe other will be responsible for the treatment phase:Treatment for Temporomandibular Disorder (TMD) and Treatment Oculomotor plus Treatment for TMD. A third-party collaborator will process and statistically analyze the collected data.Individuals will be randomize using the statistical program, two groups.Randomization and concealment of allocation will be made by a fourth external employee,not a research participant, who will organize the allocation in individual opaque envelopes and keep it confidential.There will be 2 blocks of 25 envelopes:Treatment for TMD and Treatment Oculomotor plus Treatment for TMD.With this process, participants will have the same probability of being allocated to one of the two treatment groups.Blinding of the evaluator will be maintained until the end of the research and data tabulation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oculomotor Therapy (Experimental): The procedures for oculomotor therapy will be arranged sequentially, from easiest to most difficult. It will consist of a convergence technique (Brock Cord and Barrille Cartouche) and an accommodative technique (Eccentric circles or lifesaving cards) and Eye Relaxation.
  Interventions: Other: Oculomotor Therapy
- Therapy for Temporomandibular Disorder (Active Comparator): Extra-oral and intra-oral massage: The main objective is to reduce pain as well as re-establish proper muscle length and flexibility. The patient will be instructed to use diaphragmatic breathing to promote relaxation during these massage procedures.
  Myofascial release of the masseter, temporalis and sternocleidomastoid muscles, release of neck soft tissues, cervical pomp, suboccipital inhibition, passive anteroposterior mobilization of the upper cervical, cervical exercises, Temporomandibular Joint exercises (mouth opening exercise with tongue on palate) , Proprioceptive exercises).
  Interventions: Other: Oculomotor Therapy; Other: Therapy for Temporomandibular Disorder

INTERVENTIONS:
Other: Oculomotor Therapy — It will consist exercise of a convergence technique and an accommodative technique.
Other: Therapy for Temporomandibular Disorder — It will consist exercise of a ATM and cervical spine.
  Arms: Therapy for Temporomandibular Disorder

SUMMARY:
Temporomandibular Disorder is a disorder that involves the muscles of mastication, the temporomandibular joint (TMJ), and associated structures. Convergence insufficiency (CI) is characterized by the inability of the eyes to perform the eye adduction movement together, to focus on a nearby object. Studies show that there is a relationship between the presence of TMD and its signs and symptoms in patients with convergence insufficiency. Given this, the research question of this clinical trial is whether the effect of oculomotor therapy would be effective in improving the signs and symptoms of Temporomandibular Disorder. The design of this research is a Clinical Trial, Randomized and Blind. It will be divided into two moments: evaluation and intervention. The evaluations will be carried out using the Diagnostic Criteria for Temporomandibular Disorders: Fonseca Anamnestic Index (IAF), Clinical Protocol and Assessment Instruments (DC/TMD), Mandibular function Impairment Questionnaire (MFIQ), Numerical Pain Scale (END), Convergence Test, Meersseman Test and Convergence insufficiency symptom Survey (CISS). Individuals will be randomized into 2 groups: Group A (Treatment for Temporomandibular Disorder) and Group B (Treatment Oculomotor plus Treatment for Temporomandibular Disorder). Both groups will receive physiotherapeutic treatment for 12 weeks. Patients will be reassessed shortly after treatment, 3 and 6 months later. For data analysis, the statistical significance considered will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Presence of pain in the facial region in the last 6 months;
* Presence of pain, at least 3 on the numeric pain scale (END), in the Temporomandibular Joint and/or masticatory muscles and in the last 6 months;
* Diagnosis of myogenic Temporomandibular Disorder, by DC/TMD;
* Moderate and Severe Temporomandibular Disorder carrier, according to Fonseca's Anamnestic Index;
* Presence of Insufficiency of Convergence according to Convergence Test (TC) and by Convergence insufficiency symptom Survey (CISS).

Exclusion Criteria:

* Permanent strabismus;
* History of strabismus surgery;
* History of cervical and/or craniofacial trauma/surgical procedure;
* History of ocular nerve injury;
* Neurological disorders;
* disc disease ;
* Systemic diseases;
* Fibromyalgia diagnosis;
* Previous treatments for TMD carried out in the last 3 months;
* Previous treatments of Convergence Insufficiency with oculomotor therapy (no more than 2 months of treatment in the last year);
* Occlusal treatment in progress;
* Any ocular or systemic medication known to affect accommodation or vergence ;
* Systemic diseases that affect ocular accommodation, vergence , and motility, such as multiple sclerosis, Graves' thyroid disease, myasthenia gravis, diabetes, and Parkinson's disease;
* In continuous use of analgesics, anti-inflammatories, anxiolytics and/or antidepressants;
* Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Score in Numerical Pain Scale | The level of pain at 12 weeks
  intensity of pain
Score in Numerical Pain Scale | The level of pain at 3 months
  intensity of pain

SECONDARY OUTCOMES:
measure range of motion | The range of motionat 12 weeks
  range of motion
measure range of motion | The range of motion at 3 months
  range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Daniela Aparecida Biasotto Gonzalez, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data is confi dential, but if any journal requests open data for publication for sure we will provide our database